CLINICAL TRIAL: NCT02873975
Title: A Phase II Study of the CHK1 Inhibitor LY2606368 in Patients With Advanced Solid Tumors Exhibiting Replicative Stress or Homologous Recombination Repair Deficiency
Brief Title: A Study of LY2606368 (Prexasertib) in Patients With Solid Tumors With Replicative Stress or Homologous Repair Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Geoffrey Shapiro, MD, PhD, Geoffrey Shapiro M.D., PhD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-281
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Solid tumors; MYC amplification; CCNE1 amplification; Rb loss; FBXW7 mutation; BRCA1 mutation; BRCA2 mutation; PALB2 mutation; RAD51C mutation; RAD51D mutation; ATR mutation; ATM mutation; CHK2 mutation; Fanconi anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Homologous Repair (HR) Deficiency Cohort (Experimental): Prexasertib (LY2606368) will be administered as an IV infusion in patients with homologous repair (HR) deficiency on day 1 and day 15 of every 28 day cycle. Prexasertib will be given at the recommended phase 2 dose of 105 mg/m2 administered over approximately 1 hour.
  Interventions: Drug: LY2606368
- Replicative Stress Cohort (Experimental): Prexasertib (LY2606368) will be administered as an IV infusion in patients with advanced solid tumors exhibiting replicative stress on day 1 and day 15 of every 28 day cycle. Prexasertib will be given at the recommended phase 2 dose of 105 mg/m2 administered over approximately 1 hour.
  Interventions: Drug: LY2606368
- CCNE1 Amplification Cohort (Experimental): Prexasertib (LY2606368) will be administered as an IV infusion in patients with CCNE1 amplification on day 1 and day 15 of every 28 day cycle. Prexasertib will be given at the recommended phase 2 dose of 105 mg/m2 administered over approximately 1 hour.
  Interventions: Drug: LY2606368

INTERVENTIONS:
Drug: LY2606368
  Other Names: Prexasertib

SUMMARY:
This research study is studying a checkpoint kinase 1 (CHK1) inhibitor as a possible treatment for advanced solid tumors that harbor genetic alterations in the homologous repair (HR) pathway, genetic alterations that indicate replication stress, or with CCNE1 amplification.

DETAILED DESCRIPTION:
This is an open label, phase II, two-arm study exploring the anti-tumor activity of the CHK1 inhibitor prexasertib (LY2606368) in patients with advanced solid tumors exhibiting one of the following:

1. Replicative stress, including MYC amplification, CCNE1 amplification, Rb loss, or an FBXW7 mutation
2. An HR deficiency, including tumors with genomic or somatic mutations of BRCA1, BRCA2, PALB2, RAD51C, RAD51D, ATR, ATM, CHK2, or the Fanconi anemia pathway genes
3. A CCNE1 amplification

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a pathologically confirmed advanced solid tumor for which standard therapy proven to provide clinical benefit does not exist or is no longer effective.
* Participants must have one of the following (confirmed via targeted NextGeneration sequencing [NGS] using the DFCI/BWH OncoPanel or another CLIA-certified method):

  * For the replicative stress cohort: MYC amplification, CCNE1 amplification, Rb loss, FBXW7 mutation, or another genomic abnormality indicative of replicative stress as agreed upon with the principal investigator. OR
  * For the HR deficiency cohort: genomic or somatic mutation in BRCA1, BRCA2, PALB2, RAD51C, RAD51D, ATR, ATM, CHK2, the Fanconi anemia pathway genes, or another genomic or somatic mutation in a known HR gene as agreed upon with the principal investigator.
  * For the CCNE1 cohort: CCNE1 amplification of 6-fold or greater. Patients with borderline amplification levels may be considered following approval from the overall principal investigator.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Age ≥ 18 years.
* ECOG performance status < 2
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/uL
  * Platelet count ≥ 100 K/uL
  * Hemoglobin ≥ 9 g/dL (with or without transfusion support)
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN, unless liver metastases are present and then ≤ 5 × institutional ULN is acceptable
  * Serum creatinine ≤ 1.5 × institutional ULN
* Participants enrolling to the HR or replicative stress cohorts during Stage 1 must have disease that is amenable to biopsy and be willing to undergo a pre-treatment tumor biopsy.
* The potential effects of LY2606368 use during pregnancy and lactation are not known. Nonclinical studies of LY2606368 on pregnancy and fetal development have not been performed. To minimize any potential risks, men and women with reproductive potential should use medically approved contraceptive precautions during treatment and for 3 months following the last dose of LY2606368. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 3 months after completion of LY2606368 administration.
* Ability to understand and the willingness to sign a written informed consent document.
* QTcF value of ≤ 470 msec on screening electrocardiogram (EKG)

Exclusion Criteria:

* Participants who have had chemotherapy, other investigational or biologic therapy, major surgery, or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the planned first dose of LY2606368 therapy.
* Participants who have not recovered to eligibility levels from prior toxicity or adverse events as a result of previous treatment prior to the study.
* Participants who have received prior treatment with a CHK1 inhibitor.
* Participants who have received prior radiation therapy to > 25% of the bone marrow.
* Participants with known untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with a history of brain metastases that have been treated, are no longer taking corticosteroids, and have been stable on imaging for at least one month following the end of treatment are permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LY2606368.
* Participants with a personal or family history of long QT syndrome.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, NYHA Class III/IV heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction within 3 months of enrollment, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding females. The potential effects of LY2606368 use during pregnancy and breastfeeding are not known and LY2606368 has the potential for teratogenic or abortifacient effects.
* Known HIV-positive participants are ineligible because these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in HIV-positive participants when indicated.
* Participants enrolling to the HR or replicative stress cohort during Stage 1 may not be on anticoagulant therapy unless the treating investigator has deemed it safe to temporarily hold to facilitate the pre-treatment tumor biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Homologous Repair (HR) Deficiency Cohort: Prexasertib (LY2606368) will be administered as an IV infusion in patients with homologous repair (HR) deficiency on day 1 and day 15 of every 28 day cycle. Prexasertib will be given at the recommended phase 2 dose of 105 mg/m2 administered over approximately 1 hour.
  LY2606368
- Replicative Stress Cohort: Prexasertib (LY2606368) will be administered as an IV infusion in patients with advanced solid tumors exhibiting replicative stress on day 1 and day 15 of every 28 day cycle. Prexasertib will be given at the recommended phase 2 dose of 105 mg/m2 administered over approximately 1 hour.
  LY2606368
- CCNE1 Amplification Cohort: Prexasertib (LY2606368) will be administered as an IV infusion in patients with CCNE1 amplification on day 1 and day 15 of every 28 day cycle. Prexasertib will be given at the recommended phase 2 dose of 105 mg/m2 administered over approximately 1 hour.
  LY2606368
Period: Overall Study
Arm/Group | Homologous Repair (HR) Deficiency Cohort | Replicative Stress Cohort | CCNE1 Amplification Cohort
Started | 8 | 10 | 9
Completed | 8 | 10 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Homologous Repair (HR) Deficiency Cohort | Replicative Stress Cohort | CCNE1 Amplification Cohort | Total
Number analyzed (Participants) | 8 | 10 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (9.5) | 55.2 (14.2) | 61.2 (11.6) | 59.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 13
  Male | 3 | 7 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 8 | 10 | 9 | 27
  Hispanic | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Rate at 4 Month
Description: Progression-Free Rate defines as the percentage of participants progression-free at 4 months in all arms, by RECIST 1.1 criteria. Progression-free rate will be estimated as binomial proportion and overall survival and progression-free survival estimates and curves will be generated using the Kaplan-Meier method.
Time Frame: at 4 month
Measure: Number; unit: percentage of participants
Arm/Group | Homologous Repair (HR) Deficiency Cohort | Replicative Stress Cohort | CCNE1 Amplification Cohort
Number analyzed (Participants) | 8 | 10 | 9
percentage of participants
  >= 4 months | 25 | 10 | 44.4
  < 4 months | 75 | 90 | 55.6

2. Secondary Outcome: Incidence of Grade 4 Treatment-Related Toxicity
Description: All grade 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEvE as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 4 AE of any type during the time of observation.
Time Frame: Assessed cycle 1 at day 1, 8, 15 and 22, and cycle 2 at day 1 and 15, from time of first dose and up to day 30 post-treatment. Median treatment duration for this study cohort was 55 day (range 6 - 539 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Homologous Repair (HR) Deficiency Cohort | Replicative Stress Cohort | CCNE1 Amplification Cohort
Number analyzed (Participants) | 8 | 10 | 9
Participants | 5 | 7 | 7

3. Secondary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and on treatment; Treatment continued until disease progression or unacceptable toxicity. Median treatment duration for this study cohort was 55 day (range 6 - 539 days).
Measure: Number; unit: proportion of participant
Arm/Group | Homologous Repair (HR) Deficiency Cohort | Replicative Stress Cohort | CCNE1 Amplification Cohort
Number analyzed (Participants) | 8 | 10 | 9
proportion of participant | 0 | 0 | 0.11

4. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Participants were followed long-term for survival months from the end of treatment until death or lost to follow-up. Median (range) follow-up was 133 days (15-862 days) in this study cohort.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Homologous Repair (HR) Deficiency Cohort | Replicative Stress Cohort | CCNE1 Amplification Cohort
Number analyzed (Participants) | 8 | 10 | 9
days | 108 [15 to 239] | 328 [22 to 690] | 165 [123 to 724]

ADVERSE EVENTS:
Time Frame: Assessed cycle 1 at day 1, 8, 15 and 22, and cycle 2 at day 1 and 15, from time of first dose and up to day 30 post-treatment. Median treatment duration for this study cohort was 55 day (range 6 - 539 days).
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Homologous Repair (HR) Deficiency Cohort | Replicative Stress Cohort | CCNE1 Amplification Cohort
All-Cause Mortality (participants affected / at risk) | 2/8 | 2/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 8/8 | 7/10 | 9/9
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Homologous Repair (HR) Deficiency Cohort (N=8) | Replicative Stress Cohort (N=10) | CCNE1 Amplification Cohort (N=9)
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 8 | 7 | 9
Platelet count decreased (Investigations) | 4 | 2 | 4
Sepsis (Infections and infestations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 6 | 6 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Homologous Repair (HR) Deficiency Cohort (N=8) | Replicative Stress Cohort (N=10) | CCNE1 Amplification Cohort (N=9)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0
Alkaline phosphatase increased (Investigations) | 3 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 7 | 8 | 8
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 5 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 2 | 1 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 1
Fatigue (General disorders) | 6 | 0 | 0
Fever (General disorders) | 5 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 6 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 4 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
White blood cell decreased (Investigations) | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT02873975/Prot_SAP_000.pdf